CLINICAL TRIAL: NCT06359236
Title: Bilişsel Davranışçı Terapi Temelli Kilo Kontrolü Mobil "Bİ'KİLO" Uygulamasının Geliştirilmesi ve Etkililiğinin Sınanması
Brief Title: Development and Effectiveness of Cognitive Behavioral Therapy Based Weight Control Mobile Application "BI'KILO"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ali Ercan Altinoz, Assoc. Prof. of Psychiatry, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122S049
Record Dates: First submitted 2024-03-06; First posted 2024-04-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss; Obesity; Overweight and Obesity; Eating Behavior; Eating Habit
Keywords: cognitive behavioral therapy; e-health applications; obesity; weight control
MeSH Terms: conditions — Weight Loss; Obesity; Overweight; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group will be involved in a process that includes three phases of the study: preparation phase, implementation phase and follow-up phase.
  Interventions: Other: BI'KILO Intervention
- Control Group (No Intervention): The control group will not be able to access the entire treatment program content. However, they will be able to access animation contents such as energy balance training, eating change, planning where and when and what to eat, healthy weight loss targets, three main and three snacks, determining weight loss targets and informational content titled diet types specified in the nutrition education module for a period of 6 weeks.

INTERVENTIONS:
Other: BI'KILO Intervention — The study consists of three stages: preparation phase, implementation phase and follow-up phase. During the preparation phase, participants' weight and body fat ratio will be calculated using a body analysis scale, and their height, waist and hip circumference will be measured.
  The implementation phase will last six weeks and consists of six modules, each lasting one week. The skills and practices aimed to be acquired in each module will be required to be applied in the following practice modules.
  At the end of the implementation phase, participants' weight, waist and hip circumferences will be measured again.
  The final phase, called the follow-up phase, will last four weeks. During this phase, participants will continue to keep a self-monitoring record of their eating and physical exercise, complete a hunger scale, and application card notifications will continue to be displayed.
  Arms: Treatment Group

SUMMARY:
The primary purpose of this project is to observe the effects of Cognitive Behavioral Psychotherapy-based weight-loss mobile application (Bi' Kilo) in 4 essential areas (Anthropometric, Biochemical, Psychometric, Cognitive) in overweight and obese individuals and to test whether these effects will persist after ten weeks. In this context, the original value of the proposed study is that a mobile application will be produced that is suitable for the culture and whose effectiveness has been scientifically proven.

In our current project proposal, the measurements of the participants will be evaluated holistically together with both tests and inventories, as well as physical measurements and biochemical data. In this study, the usability of the mobile application to be developed will also be evaluated and reported.

The study group of the research will consist of overweight and obese individuals. The first stage will be a pilot study to identify the shortcomings of the Bi'Kilo mobile application. After eliminating the deficiencies of the Bi' Kilo mobile application, a working group will be formed in the second phase of the research. At this stage, the sample will be divided into two different groups within the scope of the study and a study group and a control group will be formed.

The study consists of three phases as preparation, implementation, and follow-up. Measurements of the participants will be made at the beginning (Anthropometric, Biochemical, Psychometric, Cognitive), at the end of the six-week implementation phase (Anthropometric), and at the end of the four-week follow-up phase (Anthropometric, Biochemical, Psychometric, Cognitive).

DETAILED DESCRIPTION:
The primary purpose of this project is to observe the effects of Cognitive Behavioral Psychotherapy-based weight-loss mobile application (Bi' Kilo) in 4 essential areas (Anthropometric, Biochemical, Psychometric, Cognitive) in overweight and obese individuals and to test whether these effects will persist after ten weeks.

In this context, the original value of the proposed study is that a mobile application will be produced that is suitable for the culture and whose effectiveness has been scientifically proven. In the studies in the literature, obesity assessment is evaluated with anthropometric data. However, the evaluation of biochemical data in studies is limited. In our current project proposal, the measurements of the participants will be evaluated holistically together with both tests and inventories, as well as physical measurements and biochemical data. Furthermore, the usability of any application developed in the literature has not been evaluated. Usability is a crucial variable for mobile apps and web pages. In this study, the usability of the mobile application to be developed will also be evaluated and reported. Thus, an application that can be used as well as effective will be revealed.

The study group of the research will consist of overweight and obese individuals. The first stage will be a pilot study to identify the shortcomings of the Bi'Kilo mobile application. After eliminating the deficiencies of the Bi' Kilo mobile application, a working group will be formed in the second phase of the research. At this stage, the sample will be divided into two different groups within the scope of the study and a study group and a control group will be formed. The minimum sample size of the study was adopted as 70, and it is aimed to be completed with a minimum of 38 people, taking into account possible dropouts.

The study consists of three phases as preparation, implementation, and follow-up. Measurements of the participants will be made at the beginning (Anthropometric, Biochemical, Psychometric, Cognitive), at the end of the six-week implementation phase (Anthropometric), and at the end of the four-week follow-up phase (Anthropometric, Biochemical, Psychometric, Cognitive).

Within the scope of this project, it is stated that by using the Bi' Kilo mobile application, weight loss and reduction in body mass index value can be achieved in overweight and obese individuals; it is possible to reduce the HOMA-IR score, which shows insulin resistance and is a significant health problem in these individuals; it is possible to improve the hormone values indirectly related to obesity, such as leptin and ghrelin, and to improve the eating attitudes and behaviors of individuals; It is predicted that cognitive skills such as risk adjustment, impulsivity and decision making can be improved.

With this project;

1. Gaining healthy eating and active living habits and measuring its change with a 10-week practice,
2. Due to the increase in the frequency of use of the mobile application, which is supported by scientific data and prepared in accordance with our language and culture, due to geographical, economic, cultural, and social stigma factors, we do not provide weight control service. Providing equal opportunity for individuals who cannot afford this service and increasing the fight against obesity-excess weight
3. Thus, prevention of increased health expenditures and loss of workforce due to obesity and overweight It is thought that with the mobile application to be developed within the scope of the research, a product that can be used all over the country will be revealed, and this product can be made into a commercial product that can be purchased individually. With the research findings, it is planned to publish two international research articles, two international papers, and a medical specialization thesis. Furthermore, the study's findings will pave the way for the development of applications for problem areas in new graduate theses on the production of self-help content in different fields.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study
* being literate
* being overweight
* being over the age of 18

Exclusion Criteria:

* Being diagnosed with substance and/or alcohol use disorder
* being illiterate
* Being pregnant or having a pregnancy plan during the research period
* Being diagnosed with a disease that causes neuroendocrine obesity (Cushing's disease, hypothyroidism, hypothalamic obesity, growth hormone deficiency, hypogonadism, pseudohypoparathyroidism, polycystic ovary syndrome)
* Using antipsychotics, antiobesity drugs or cortisone-containing drugs
* Being a cigarette-smoker
* If the participant withdraws his/her consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Body Mass Index is a person's weight in kilograms divided by the square of height in meters.

SECONDARY OUTCOMES:
Weight | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  The value of body weight in kilograms.
Height | Pre-test
  The value of a person's height in centimeters.
Waist Circumference (WC) | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Waist circumference is measured halfway between the lower ribs and the iliac crest, while hip circumference is measured at the largest circumference around the buttocks.
Hip Circumference | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  The distance around the human body at the level of maximum posterior extension of the buttocks.
Waist-Hip Ratio (WHR) | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement.
Body Fat Percentage (BFP) | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Body fat percentage (BFP) is a person's total fat mass divided by total body mass multiplied by 100; body fat includes essential body fat and stored body fat. Body fat percentage will be measured using a body analysis scale.
Visceral Fat | Pre-test, post-test (6 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Visceral fat is belly fat found deep within person's abdominal cavity. Visceral fat will be measured using a body analysis scale.
Blood Glucose Level | Pre-test, follow up (10 weeks later from pre-test)
  The measure of glucose concentrated in the blood. At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes. Blood glucose level measurements will be made from the separated serums.
Blood Insulin Level | Pre-test, follow up (10 weeks later from pre-test)
  A hormone made by the islet cells of the pancreas. At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes. Blood insulin level measurements will be made from the separated serums.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Pre-test, follow up (10 weeks later from pre-test)
  Homeostasis model assessment of insulin resistance (HOMA-IR) is a method to measure insulin resistance. HOMA-IR score will be calculated as Fasting Glucose (mg/dL) X Fasting Insulin (uIU/mL) /405.
Serum Leptin Level | Pre-test, follow up (10 weeks later from pre-test)
  Leptin is an adipocyte-derived hormone and has shown positive correlation with obesity and metabolic syndrome (MetS). At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes. The remaining serum will be stored at -80°C, and Leptin levels will be studied from these stored samples.
Serum Ghrelin Level | Pre-test, follow up (10 weeks later from pre-test)
  Ghrelin is an orexigenic peptide predominantly secreted from the stomach and stimulates appetite and growth hormone release. At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes. The remaining serum will be stored at -80°C, and Ghrelin levels will be studied from these stored samples.
Emotional Eating Scale (EES) Turkish Form | Pre-test, follow up (10 weeks later from pre-test)
  The scale is a Likert-type scale consisting of 30 items, developed by Bilgen et al. and whose validity and reliability study was conducted (Bilgen, 2018). Developed as a result of the findings obtained from validity and reliability studies, TEES consists of 30 items expressing eating behavior in positive and negative emotions and includes 4 subtypes: Eating in situations of tension, eating to cope with negative emotions, self-control, control over stimuli.
Mindful Eating Questionnaire (MEQ) Turkish Form | Pre-test, follow up (10 weeks later from pre-test)
  The validity and reliability study of the Turkey form was conducted by Köse et al. in 2016 (Köse, Tayfur, Birincioğlu, & Dönmez, 2016). The Eating Awareness Scale, which consists of 30 Likert-type questions, includes 7 subtypes: eating without thinking, emotional eating, eating control, awareness, eating discipline, conscious nutrition, being affected by external factors.
Modified Yale Food Addiction Scale Version 2.0 Turkish Form (mYFAS 2.0) | Pre-test, follow up (10 weeks later from pre-test)
  The Yale Food Addiction Scale (YFAS) operationalizes indicators of addictive-like eating, originally based on the Diagnostic and Statistical Manual of Mental Disorders 4th edition Text Revision (DSM-IV-TR) criteria for substance-use disorders. The YFAS has multiple adaptations, including a briefer scale (mYFAS). Recently, the YFAS 2.0 was developed to reflect changes to diagnostic criteria in the DSM-5 (Schulte 2017).
Motor Screening Task (MOT) | Pre-test, follow up (10 weeks later from pre-test)
  The Motor Screening Task provides a general assessment of whether sensorimotor deficits or lack of comprehension, will limit the collection of valid data from the participant.
Spatial Working Memory (SWM) | Pre-test, follow up (10 weeks later from pre-test)
  Spatial Working Memory Test: In this test, comprehension and management of visual-spatial information is measured. This test, which also requires the use of some executive functions, provides measurements for working memory errors and strategy determination. It is implemented through CANTAB. It takes approximately 10-12 minutes.
Stop Signal Task (SST) | Pre-test, follow up (10 weeks later from pre-test)
  In this test, response inhibition (impulse control) is measured. It is implemented through CANTAB. It takes approximately 14 minutes.
Rapid Visual Information Processing (RVP) | Pre-test, follow up (10 weeks later from pre-test)
  Developed to measure sustained attention. It is implemented through CANTAB. It takes approximately 5-9 minutes and outcome measures include response rate, false alarms, and specificity.
Cambridge Gambling Test (CGT) | Pre-test, follow up (10 weeks later from pre-test)
  This test was developed to assess decision-making and risk-taking behavior outside a learning context. It is implemented through CANTAB. The outcome measures of this test, which takes approximately 15-20 minutes, include risk taking, decision-making quality, decision time, risk adjustment, delay reluctance and impulsivity measurements.

OTHER OUTCOMES:
Demographic Information Form | Pre-test
  In this form, in addition to the participant's gender, age and education level, information such as marital status, occupation, education level, past or current use of psychiatric medication, history of psychiatric illness in family history, history of physical illness in family history, alcohol and substance use, and economic status are also gathered.
Structured Clinical Interview for DSM-5 Disorders (SCID-5) | Pre-test
  SCID-5 was developed by First et al. It consists of 10 modules. Modules include psychotic symptoms, psychotic disorders, mood disorders, substance use disorders, anxiety disorders, obsessive-compulsive disorder and related disorders, as well as post-traumatic stress disorder, attention deficit and hyperactivity disorder, probing questions for other disorders, and adjustment disorder (American Psychiatric Association 2015) . SCID-5 can be applied to individuals over the age of 18 who do not have severe cognitive deficits, severe psychotic symptoms, or agitation. Sources of information are the patient himself, the patient's family and relatives, the healthcare team, medical sources and observations. If necessary, corrections can be made in the light of additional information and can be completed in more than one session. Average application time is 40-60 minutes. Its adaptation into Turkish and its reliability were investigated by Elbir et al.
The Eating Disorder Assessment for DSM-5 (EDA-5) | Pre-test
  The EDA-5 is a semi-structured interview intended to assist in the assessment of a feeding or eating disorder or related conditions according to DSM-5 criteria. It is designed for use by clinicians (across disciplines) with some familiarity with feeding and eating disorder diagnoses. The Turkish version was adapted by Ezgi Deveci, H. Özlem Sertel Berk and Başak Yücel (Deveci, 2019).
Blood ACTH Level (ACTH) | Pre-test
  The ACTH test measures the level of adrenocorticotropic hormone (ACTH) in the blood. ACTH is a hormone released from the pituitary gland at the base of the brain. At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes.ACTH measurements will be made from the separated serums.
Blood Growth Hormone Level (GH) | Pre-test
  Growth Hormone, peptide hormone secreted by the anterior lobe of the pituitary gland. GH stimulates protein synthesis and increases fat breakdown to provide the energy necessary for tissue growth. At 08.00 in the morning, after at least 8 hours of fasting, 8 ml of blood will be collected into vacuum gel tubes with a vacuum blood collection system and after waiting for the clotting time of the blood samples, they will be centrifuged at 1500 g for 10 minutes. GH measurements will be made from the separated serums.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available on request from the corresponding author, A.E.A. The data are not publicly available due to restrictions that their containing information that could compromise the privacy of research participants.